CLINICAL TRIAL: NCT00815074
Title: Military Women's Health and Illness Behaviors in Deployed Settings
Status: Completed | Type: Observational
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Candy Wilson, Candy Wilson, PhD, APRN, WHNP-BC, FAAN, 59th Medical Wing
Other Study IDs: HU0001-08-1-TS11
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Genitourinary Symptoms
Keywords: Military Women; Women's Health; Genitourinary Symptoms; Illness Behaviors; To determine how women manage genitourinary symptoms while deployed.
MeSH Terms: conditions — Illness Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women in the military who have returned from deployment within the past 12 months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
The purpose of this study is to gain better understanding of how recently deployed military women managed urinary and vaginal symptoms while deployed. Participants in this study will be asked to take part in a 45-60 minute interview.

ELIGIBILITY:
Inclusion Criteria:

* Deployment within the last 12 months
* Managed genitourinary symptoms while deployed (does not have to be diagnosed by a medical provider)

Exclusion Criteria:

* Women who are assigned to a medical group/hospital

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 military women.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2010-12-15 (Actual); Study Completion 2011-12-15 (Actual)

PRIMARY OUTCOMES:
Description of deployed experience using qualitative methods | 2008 to 2011
  interview data analysis

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CR Darnall Army Medical Center, Fort Hood, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas

IPD SHARING:
Plan to Share IPD: No
there will be no sharing of the data. The data have been destroyed.

REFERENCES:
- [Background] Wilson C, Corrigan R, Braun L. Deployed women's illness behaviors while managing genitourinary symptoms: An exploratory theoretical synthesis of two qualitative studies. Nurs Outlook. 2017 Sep-Oct;65(5S):S17-S25. doi: 10.1016/j.outlook.2017.07.009. Epub 2017 Jul 15. PMID 28800835
- [Result] Wilson C, Nelson JP. Exploring the patterns, practices, and experiences of military women who managed genitourinary symptoms in deployed settings. J Obstet Gynecol Neonatal Nurs. 2012 Mar;41(2):293-302. doi: 10.1111/j.1552-6909.2012.01347.x. PMID 22834851